CLINICAL TRIAL: NCT05447923
Title: Colorectal Cancer Screening in Black and Underserved Communities in the Phoenix Metro Area: Addressing Disparities in Cancer Prevention
Brief Title: Addressing Disparities in Colorectal Cancer Screening in Black and Underserved Phoenix Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21-009729; NCI-2022-04529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FIT DOM (Other: Mayo Clinic Women's Health)
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (FIT, education, questionnaire, patient navigation) (Experimental): Participants receive free FIT tests in conjunction with education on colorectal cancer screening. Participants undergo self-collect FIT and mail the sample to Mayo Clinic Lab for processing. Participants also complete a questionnaire about colorectal cancer screening and healthcare. Participants receive FIT test results through Mayo Clinic nursing support and participants with a positive test are followed up by a patient navigator to discuss next steps and consultation with a gastroenterologist to review their results.
  Interventions: Other: Educational Intervention; Other: Fecal Immunochemical Test; Behavioral: Patient Navigation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Undergo education for colorectal cancer screening
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Fecal Immunochemical Test — Undergo FIT testing
  Other Names: FIT; iFOBT; immunoassay fecal occult blood test; immunochemical fecal occult blood test; Immunochemical FOBT; immunologic fecal occult blood test
Behavioral: Patient Navigation — Undergo patient navigation for positive FIT results
  Other Names: Patient Navigator Program
Other: Questionnaire Administration — Complete questionnaire about colorectal cancer screening and healthcare

SUMMARY:
This clinical trial studies disparities involving colorectal cancer prevention and screening in Black and underserved communities in the Phoenix metropolitan area. The Black community is disproportionately impacted by colorectal cancer, with the highest rate of any racial/ethnic group in the United States. There are complex reasons behind these disparities, largely related to socioeconomic factors and healthcare access. Providing access to free, home-based fecal immunochemical testing (FIT), colorectal screening education, and appropriate follow-up to predominantly Black community-based organizations and underserved communities may help to close this gap.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate patient navigation to address colorectal cancer disparities seen in people of color, minority populations, and establish an ongoing colorectal cancer screening outreach program for this community in Phoenix.

OUTLINE:

Participants receive free FIT tests in conjunction with education on colorectal cancer screening. Participants undergo self-collect FIT and mail the sample to Mayo Clinic Lab for processing. Participants also complete a questionnaire about colorectal cancer screening and healthcare. Participants receive FIT test results through Mayo Clinic nursing support and participants with a positive test are followed up by a patient navigator to discuss next steps and consultation with a gastroenterologist to review their results.

After completion of screening, participants with a positive FIT test are followed up at 2 and 4 weeks after initial outreach to assure participants have received adequate follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years of age or older
* No prior history of colorectal cancer or colon polyps
* No first-degree family history of colorectal cancer who were diagnosed under age 60
* No current gastrointestinal (GI) or rectal symptoms (such as rectal bleeding)
* Have not undergone a colonoscopy in the last 5 years
* Have not had a fecal immunochemical test (FIT) test within the last year
* Participants that attend 4 predominantly African American churches within the Phoenix Community and extend the study opportunity as feasible to other underserved communities in the Phoenix Metro area

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer disparities seen in people of color and minority populations | Up to study completion, up to 30 days
  Evaluate patient navigation to address colorectal cancer disparities seen in people of color, minority populations, and establish an ongoing colorectal cancer screening outreach program.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana M. Kling, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials